CLINICAL TRIAL: NCT03023553
Title: The Human Mucosal Immune Responses to Influenza Virus: A Systems Biology Approach. Innate Immune Responses to Influenza Virus in Single Human Nasal Epithelial Cells
Brief Title: The Human Mucosal Immune Responses to Influenza Virus (SLVP026)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-25537; U19AI090019 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: Trivalent, inactivated influenza vaccine; Live, attenuated influenza vaccine; Nasopharyngeal swabs; Young adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIV Group (Other): Healthy adult males and females, 18-30 years of age. Immunization with standard trivalent, inactivated influenza vaccine (TIV), Fluzone®.
  Interventions: Biological: Fluzone®
- LAIV Group (Other): Healthy adult males and females, 18-30 years of age. Immunize with intranasal live, attenuated influenza vaccine (LAIV), FluMist®.
  Interventions: Biological: FluMist®

INTERVENTIONS:
Biological: Fluzone® — Influenza Virus Vaccine Suspension for Intramuscular Injection
  Arms: TIV Group
Biological: FluMist® — Influenza Virus Vaccine Live, Intranasal Spray
  Arms: LAIV Group

SUMMARY:
This study will examine the immune responses to the seasonal influenza vaccine in single cells of the nasal passages when compared with cells in circulating blood.

DETAILED DESCRIPTION:
Using state-of-the-art technology, the investigators hope the information learned from this study will help identify and describe important factors in the early-stage development of influenza immunity and possibly lead to the development of more effective vaccines. This study will be conducted in healthy male and female volunteers 18-30 years of age who received one of two seasonal influenza vaccine types, intramuscular standard trivalent inactivated influenza vaccine (TIV) or live, attenuated influenza vaccine (LAIV) given by intranasal spray.

Participants are divided into two groups. The control group will receive the 2012-2013 formulation of the standard intramuscular trivalent inactivated influenza vaccine (TIV). A blood sample and nasopharyngeal swab samples (one from each nostril) will be collected at a single visit, Day 0. For those in the live, attenuated influenza vaccine (LAIV) group, at the first visit, they will receive a single administration of the 2012-2013 formulation of LAIV. At the second study visit two days later, they will provide a blood sample and two nasopharyngeal swab samples (one from each nostril).

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, ambulatory adult between the ages of 18-30 years
2. Willing to complete the informed consent process.
3. Availability for follow-up at Day 2 (LAIV Group only)
4. Acceptable medical history by review of inclusion/exclusion criteria and vital signs.

Exclusion Criteria:

1. Prior off-study vaccination with the current 2012-2013 seasonal TIV or LAIV
2. Allergy to egg or egg products, or to vaccine components, including thimerosal (TIV multidose vials only), or gentamicin, gelatin, arginine or MSG (for LAIV only).
3. Life-threatening reactions to previous influenza vaccinations
4. Asthma or history of wheezing (except for controls in the study who will be assigned to receive TIV).
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
8. Blood pressure >150 systolic or >95 diastolic at first study visit
9. Hospitalization in the past year for congestive heart failure or emphysema.
10. Chronic Hepatitis B or C.
11. Recent or current use of immunosuppressive medication, including systemic glucocorticoids. Corticosteroid nasal sprays for allergies and topical steroids are permissible. Inhaled steroids for conditions such as asthma are not permissible for volunteers in the LAIV group.
12. Participants in close contact with anyone who has a severely weakened immune system should not receive LAIV (LAIV Group only).
13. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
14. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
15. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
16. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. aspirin per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety..
17. Receipt of blood or blood products within the past 6 months of planned used during the study.
18. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
19. Inactivated vaccine 14 days prior to vaccination or planned non-study vaccination prior to completion of the last study visit.
20. Live, attenuated vaccine within 60 days of vaccination or planned non-study vaccination prior to completion of the last study visit.
21. History of Guillain-Barré Syndrome
22. Pregnant or lactating woman
23. Use of investigational agents within 30 days prior to enrollment or planned use of investigational agents prior to completion of study visits.
24. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned donation prior to completion of the last visit.
25. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Harry Greenberg, MD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford Universityh

IPD SHARING:
Plan to Share IPD: Yes
The NIH Human Immunology Project Consortium (HIPC) data repositories (ImmPORT) may store the results of the research assays results. Genetic data that is developed in this study may be made available to other researchers through the National Center for Biotechnology Information (NCBI) databases. Results from research assays will be labeled with a unique identification code and the volunteer identity (except for age) will not be disclosed.

RESULTS

PARTICIPANT FLOW:
Groups:
- TIV/ Control Group: Healthy adult males and females, 18-30 years of age. Immunization with standard trivalent, inactivated influenza vaccine (TIV), Fluzone®.
  Fluzone®: Influenza Virus Vaccine Suspension for Intramuscular Injection
Period: Overall Study
Arm/Group | TIV/ Control Group | LAIV Group
Started | 4 | 9
Completed | 4 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: In LAIV Group, 13 subjects initially consented. One subject was determined ineligible due to age. Twelve subjects completed the LAIV Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | TIV/ Control Group | LAIV Group | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.99 (2.955) | 24.60 (5.22) | 24.40 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 8 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Each Arm Who Received Influenza Vaccine
Time Frame: Day 0 to 28
Measure: Count of Participants; unit: Participants
Arm/Group | TIV/ Control Group | LAIV Group
Number analyzed (Participants) | 4 | 9
Participants | 3 | 8

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | TIV/ Control Group | LAIV Group
Number analyzed (Participants) | 3 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 to 28
Description: Clinical Assessment performed at each visit
Arm/Group | TIV/ Control Group | LAIV Group
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/8
Other Adverse Events (participants affected / at risk) | 0/3 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No